CLINICAL TRIAL: NCT05807321
Title: Fecobionics to Monitor and Predict Biofeedback Therapy in Dyssynergia Patients
Brief Title: Fecobionics in Biofeedback Therapy in Dyssynergia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The California Medical Innovations Institute, Inc. (Other)
Collaborators: Scripps Clinic (Other); Augusta University Medical Center (Unknown)
Responsible Party: Principal Investigator, Hans Gregersen, PhD, CEO, The California Medical Innovations Institute, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CALM-CLIN-2023 BFT
Record Dates: First submitted 2023-03-16; First posted 2023-04-11 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Dyssynergia; Constipation
Keywords: Fecobionics; Biofeedback therapy; Defecation
MeSH Terms: conditions — Ataxia; Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fecobionics (Experimental)
  Interventions: Device: Fecobionics

INTERVENTIONS:
Device: Fecobionics — Fecobionics is a novel device to be inserted through the anal canal into rectum for studying defecation. Anorectal manometry and balloon expulsion test may be used as reference. Anorectal manometry and balloon expulsive test are standard methods for anorectal functional measurement.
  Other Names: Anorectal manometry; Balloon expulsive test

SUMMARY:
Constipation affects 12-19% of Americans. Pelvic floor dyssynergia is considered to play an important role in constipation but the underlying mechanisms are not well understood in individual patients. The investigators have developed a novel device named Fecobionics that provide detailed mapping of physiological parameters during defecation. The aim of the study is to use Fecobionics to assess anorectal function in dyssynergia patients and monitor and predict the outcome of the biofeedback therapy.

DETAILED DESCRIPTION:
This study aims to monitor and predict biofeedback therapy based on mechanism-based and highly integrated data using a new medical device. This study is specifically for patients with dyssynergia before, during, and after biofeedback therapy. The balloon-like Fecobionics device (10 cm long and 1 cm in diameter) will be inserted into the participant's rectum and will record data before and during the expulsion of the device. The participant will be asked to do different motions like cough, squeeze, or push during the procedure. The novel data obtained in this study may help the investigators to identify the patients who will benefit or not benefit from biofeedback therapy before the therapy is done. This will determine the effectiveness of treatments for anorectal disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent.
2. Age between 21-75 years.
3. Subjects must fulfill the criteria for obstructed defecation/dyssynergia and enter the BFT at UCSD or Scripps.

Exclusion Criteria:

1. Female who is pregnant or lactating.
2. Prior abdominal or anorectal surgery or bowel resection.
3. Diagnosis of fecal incontinence, any anorectal symptoms and drug use that affect anorectal function.
4. Confirmed or suspected COVID-19 infection.
5. Severe cardiovascular disease.
6. Subjects not willing to consent and undergo the specified tests in this study.
7. Other exclusions, that in the opinion of the investigator, the volunteer is not a suitable subject for the study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Expulsion Duration | 1.5 year
  The time it takes to defecate Fecobionics
Pressure Difference between front and rear ends of Fecobionics | 1.5 year
  A measure of anal sphincter pressure, the driving rectal pressure, and the difference between these two pressures. This is the key to the determination of defecation phases.

SECONDARY OUTCOMES:
Anorectal angle | 1.5 year
  Anorectal angle is an important parameter for defecation
Mechanical Tension of Fecobionics | 1.5 year
  To reflect anorectal function, the mechanical tension will be computed. The tension is equal to anorectal radius multiply pressure.
Expulsion Velocity | 1.5 year
  Measured from the time difference between multiple sensor data
Cross-sectional area | 1.5 year
  Computed by diameter

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - California Medical Innovations Institute, San Diego, California
  - Digestive Health Center- Augusta University, Augusta, Georgia